CLINICAL TRIAL: NCT03319134
Title: Investigating the Neural Correlates in Memory Retrieval After HD-tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Sven Vanneste, Associate professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18-01
Record Dates: First submitted 2017-10-18; First posted 2017-10-24 (Actual); Results first posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Healthy Adults

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three groups: (1) active HD-tDCS with retrieval memory task, (2) sham HD-tDCS with retrieval memory task, (3) active cathodal HD-tDCS with retrieval memory task
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- active anodal HD-tDCS (Experimental): Active anodal HD-tDCS stimulation applied during memory task
  Interventions: Device: active anodal HD-tDCS
- sham HD-tDCS (Sham Comparator): Sham HD-tDCS stimulation during memory task for comparison
  Interventions: Device: sham HD-tDCS
- active cathodal HD-tDCS (Experimental): Active cathodal HD-tDCS stimulation applied during memory task
  Interventions: Device: active cathodal HD-tDCS

INTERVENTIONS:
Device: active anodal HD-tDCS — 1) active anodal HD-tDCS with memory task
  Arms: active anodal HD-tDCS
Device: sham HD-tDCS — 2) sham HD-tDCS with memory task
  Arms: sham HD-tDCS
Device: active cathodal HD-tDCS — 3) active cathodal HD-tDCS with memory task
  Arms: active cathodal HD-tDCS

SUMMARY:
The overall objective of this study is to investigate the neural correlate in retrieval memory task.

The aim of the study is to understand the undergoing changes in late positive ERP component during retrieval memory task when stimulating the posterior cingulate cortex (PCC) with High Definition Transcranial Direct Current Stimulation (HD-tDCS).

DETAILED DESCRIPTION:
Retrieval memory is supported by distinct retrieval process known as recollection and familiarity. These two process have been associated with distinct event related potentials (ERPs). At the time of retrieval, familiarity is associated with modulation of the FN400, an enhanced positivity for old items relative to new items observed from approximately 400-600ms post stimulus onset. The FN400 tends to have mid-frontal scalp distribution which can extend to left and right frontal areas and central midline regions. In contrast, recollection has been linked with modulation of positive going waveform that emerges approximately 600ms post stimulus and is typically maximal over parietal sites and referred to as late positive component (LPC). In addition, FN400 is found to increase gradually as a function of item retrieval confidence whereas LPC is limited to high confidence retrieval response.

High Definition transcranial Direct Current Stimulation (HD-tDCS ) is a non-invasive neuromodulation technique. Compared to the standard bipolar montage used by the conventional tDCS, it uses arrays of smaller, specially designed electrodes to deliver a constant and low current directly to the cortical brain areas to increase the spatial focality. Studies show that the cortical area undergoing stimulation with HD-tDCS is more restricted compared to the standard bipolar montage of conventional tDCS. Moreover, tDCS has been proposed as a therapeutic procedure in various diseases and tDCS in healthy adults have demonstrated to improve cognitive and memory performance, but information regarding the effects of HD-tDCS targeting the PCC and its impact on memory retrieval is scarce. By targeting the PCC area by HD-tDCS, we want to introduce a safer, easier-to-use and more accurate non-invasive neuromodulation procedure. The dysfunctions of posterior cingulate cortex hav been linked to a range of psychiatric and neurological condition such as Alzheimer's disease, schizophrenia, autism, depression and attention deficit hyperactivity disorder, as well as aging. It shows increased activity when subject retrieve autobiographical memories suggests its internal orientated function. PET and ERP combined studies have shown greater blood flow medial temporal lobe with a brief late positive ERP component in PCC. Therefore, in this study we aim to understand whether HD-tDCS targeting the PCC can modulate the late positive ERP component.

ELIGIBILITY:
Inclusion Criteria:

* Native English Speaker
* Currently not using any medication
* Capable of understanding and signing an informed consent

Exclusion Criteria:

* Severe disease
* Mental illness
* Cardiac history
* History of severe head injuries
* History of epileptic seizures
* Any implanted devices such as pacemaker, neurostimulator
* Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Vanneste, Principal Investigator — The University of Texas at Dallas
Locations (1):
- University of Texas at Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Anodal HD-tDCS | Sham HD-tDCS | Active Cathodal HD-tDCS
Started | 15 | 15 | 15
Completed | 15 | 15 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Anodal HD-tDCS | Sham HD-tDCS | Active Cathodal HD-tDCS | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 45
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.8 (1.78) | 18.8 (1.32) | 18.9 (1.53) | 18.84 (1.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 11 | 33
  Male | 5 | 3 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 15 | 15 | 15 | 45
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Recognition Memory Assessed by a Retrieval Memory Experiment
Description: Participants had to learn an association between a face and a name. The face-name association memory task was divided into (1) an encoding phase, (2) a consolidation phase, and (3) a retrieval phase. During the encoding phase, participants studied 60 successively presented face-name pairs. Participants were instructed to assess the gender of each face shown to keep participants focused on the task. The encoding phase lasted approximately 5 minutes. This is followed by a consolidation phase where participants were instructed to "sit still, relax, and think about nothing in particular" for 10 minutes. During the retrieval phase, participants were presented with 60 old and 60 new faces and were instructed to assess whether they had seen this face during the encoding phase, or if it was a 'new' face. Participants received active or sham transcranial direct current stimulation targetting the posterior cingulate cortex during retrieval. The outcome is correctly recalled old faces.
Time Frame: Retrieval Memory is assessed after 90 seconds break following the recognition phase.
Measure: Mean (Standard Error); unit: percentage of correctly recalled old fac
Arm/Group | Active Anodal HD-tDCS | Sham HD-tDCS | Active Cathodal HD-tDCS
Number analyzed (Participants) | 15 | 15 | 15
percentage of correctly recalled old fac | 48.47 (4.038) | 34.78 (4.038) | 33.983 (4.662)

ADVERSE EVENTS:
Time Frame: two weeks
Description: All groups received one HD-tES procedure followed by a questionnaire about their HD-tES experience. The questionnaire was based on the tES adverse effects questionnaire proposed (Brunoni et al., 2011).
Arm/Group | Active Anodal HD-tDCS | Sham HD-tDCS | Active Cathodal HD-tDCS
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol: Study Protocol (2016-01-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT03319134/Prot_001.pdf